CLINICAL TRIAL: NCT00998530
Title: Trichomoniasis: Genotype and Phenotype Correlations in African American Women
Status: Completed | Type: Observational
Sponsor: University of Mississippi Medical Center (Other)
Collaborators: Mississippi State Department of Health (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2009-0138
Record Dates: First submitted 2009-10-13; First posted 2009-10-20 (Estimated); Last update posted 2019-05-23 (Actual); Status verified 2019-04

CONDITIONS: Trichomonas Infections
Keywords: Trichomonas vaginalis; trichomoniasis; MLST; Multilocus sequence typing
MeSH Terms: conditions — Trichomonas Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Trichomonas vaginalis clinical isolates
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- African American HIV+: African American women with HIV and infected with Trichomonas
- Caucasian HIV-: Caucasian women who are HIV negative and infected with Trichomonas
- African American HIV-: African American women who are HIV negative and are infected with Trichomonas

SUMMARY:
The hypothesis to be tested in this trial is that the different epidemiologic (including racial differences) and phenotypic manifestations exhibited by Trichomonas clinical isolates during infection are correlated with their genotypic strain classification. Two specific aims are proposed to test that hypothesis. Specific aim 1. Assess the significance of genotypic or phenotypic differences in the Trichomonas strains among African American women by HIV status. Specific aim 2. Determine the significance of genotypic or phenotypic differences in the Trichomonas strains circulating among women from two different racial groups, African American women and Caucasian women. The overall goals of these specific aims are to identify racial differences in the genotypic and phenotypic characteristics of Trichomonas strains, and to develop the ability to identify and classify Trichomonas infections in order to prioritize treatment and epidemiologic follow-up of individuals infected with isolates associated with adverse clinical outcomes (HIV transmission or acquisition, pregnancy complications, virulence, or drug resistance).

DETAILED DESCRIPTION:
Despite serious public health consequences, its widespread prevalence, rising drug resistance and treatment failures, little has been done to study the role of T. vaginalis genotype in transmission, virulence, occurrence of mixed infections, and the spread of drug resistance, primarily due to the lack of suitable assays for rapid strain typing. Previously utilized genotyping techniques for Trichomonas are inadequate due to problems with speed of analysis, sensitivity, and reproducibility between different labs. Multilocus sequence typing (MLST) combines speed, sensitivity, portability, accuracy, and reliability by determining nucleotide sequence polymorphisms (SNPs) present in small DNA fragments (300-400 nt) that are amplified by polymerase chain reaction (PCR) from a number (usually 6-7) of neutrally selected housekeeping genes. MLST assigns an allele fragment number (AFN) for each unique SNP or combination of SNPs present in a gene fragment and uses these to identify unique sequence types (STs) based on the AFN combinations in the collection of all the genes analyzed. MLST has been used extensively to study epidemiology, population structure, virulence and evolution in pathogenic bacteria but only for fungi among eukaryotes, due to the difficulty of interpreting MLST data in diploid organisms. However, T. vaginalis differs from other eukaryotes, possessing a stable haploid set of six chromosomes, and the investigators have developed an MLST genotyping system for T. vaginalis clinical isolates. The data (AFNs and STs) generated for each T. vaginalis strain by the MLST scheme we develop will be deposited in a freely accessible internet database. This MLST scheme will then be used to examine the relationships between strain genotypes and the clinical, epidemiologic, and physiologic manifestations of trichomoniasis.

Trichomoniasis is characterized by a wide spectrum of clinical presentation and disease sequelae. This clinical variability is accompanied by a high degree of genetic diversity in Trichomonas vaginalis clinical isolates as we originally demonstrated and others have confirmed. The investigators hypothesize that correlations between genotype and clinical presentation are true for trichomoniasis and that T. vaginalis isolates differ in their capacity for clinical disease, severity, drug resistance, and disease sequelae. In support, several studies (10-40 patients) show a statistically significant correlation between the genetic relatedness of T. vaginalis isolates, using a random amplified polymorphic DNA (RAPD) technique, with their clinical presentation. Correlations between disease severity in trichomoniasis and in vitro phenotypic properties such as cytoadherence, cytotoxicity and expression of cysteine proteinase 30 kilo-dalton (kDa) protein have also been reported. Significant differences in cytoadherence to cell monolayers, differential protein expression, phagocytosis of target cells, ability to exert cytotoxic damage on cultured cells, and pathogenicity and mortality in mice have been demonstrated in T. vaginalis clinical isolates, indicating the wide variation in virulence properties present in Trichomonas isolates. The investigators have also demonstrated up to four-fold differences in secreted cysteine protease activity between cultured T. vaginalis clinical isolates. The accumulated evidence strongly supports a correlation between individual T. vaginalis strains and their capacity for virulence.

For this specific study, at the initial enrollment/diagnosis visit the investigators will collect T. vaginalis isolates accompanied by a detailed clinical assessment, epidemiological information, and the results of in vitro testing of drug .resistance. This information will allow the investigators to determine if particular strains or groups of strains (as determined by MLST genotyping) are associated with asymptomatic infection, clinical severity, patient race, treatment failures, drug resistance, mixed infections or sexual history using univariate and multivariate analysis. This is significant because positive associations of particular strains or groups of strains with these factors, as the investigators expect to find, will necessitate changes in the way trichomoniasis is managed and treated with reference to the strains identified. The investigators will also independently test these variables for correlations with each other to identify variables or combinations of variables which may be associated with clinical manifestations of trichomoniasis.

The information the investigators gather will also permit a better understanding of trichomoniasis in many additional ways. The investigators will culture T. vaginalis at test of cure (TOC) follow-up visits to genotype and determine their drug resistance in order to distinguish potential treatment failures or conversion to drug resistance (same genotype as original visit) from re-infection by another contact (different genotype). This is particularly significant for HIV+ women as their Trichomonas vaginalis infections are more difficult to cure and T. vaginalis may persist, undetectable by culture, only to re-emerge up to six months later. Trichomonas vaginalis is detected at TOC visits at much higher rates (up to 36 %) in HIV+ women than in HIV- women (8%) with most of these infections ascribed to treatment failures. Recent reports describe persistent, undetected T. vaginalis infections cultured 3 and 6 months after an initial negative TOC result in women who report no intervening sexual contacts. This is significant as a correlation of strain genotype with persistent infection will identify HIV+ individuals needing multiple TOC visits, use of more sensitive diagnostic tests, and perhaps longer treatment courses.

ELIGIBILITY:
Inclusion Criteria:

* Trichomonas infection

Exclusion Criteria:

* pregnancy

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting to clinic sites with symptoms of a sexually transmitted disease
Sampling Method: Non-Probability Sample
Enrollment: 231 (Actual)
Dates: Start 2009-09 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Correlation of Trichomonas genotype with clinical symptoms, HIV status and patient race. | Single visit
  Trichomonas vaginalis isolates will be genotyped using Multilocus sequence typing (MLST) and the isolate genotypes will be assessed for correlations with clinical manifestations, drug resistance, HIV status, and demographic patient information.

CONTACTS AND LOCATIONS:
Overall Officials: John C Meade, PhD, Principal Investigator — University of Mississippi Medical Center
Locations (4):
- United States (4):
  - Women's Specialty Clinic at Mirror Lake, Flowood, Mississippi
  - University Physicians Grants Ferry, Flowood, Mississippi
  - Crossroads Clinics, Jackson, Mississippi
  - University Physicians Jackson Medical Mall, Jackson, Mississippi

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared with other investigators upon completion of the study and journal acceptance of manuscripts detailing study results. Data may be accessed by contacting Dr. Meade